CLINICAL TRIAL: NCT05490121
Title: Evaluating an Educational Intervention for Improving Residents' Recognition and Response to Child Maltreatment - A Mixed Method Acceptability and Feasibility Study With a Pilot Randomized Trial
Brief Title: RISE With Residents
Acronym: RISE Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Royal College of Physicians and Surgeons of Canada (Other)
Responsible Party: Principal Investigator, Melissa Kimber, PhD, MSW, RSW, Assistant Professor, Department of Psychiatry & Behavioural Neurosciences, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HiREB #14381
Record Dates: First submitted 2022-07-28; First posted 2022-08-05 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Domestic Violence; Child Maltreatment; Pediatric ALL; Psychiatry; Education, Medical, Graduate
Keywords: Family Violence; Medical Education; Education Scholarship; Health Professions Education; Mandatory Reporting; Child Maltreatment
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: To determine the feasibility of evaluating the effectiveness of both of VEGA's educational approaches, as well as to generate preliminary estimates of effect for sampling and effect size calculations, a two-arm pilot randomized controlled trial (RCT) will be used (Eldridge et al., 2016). Eligible participants will be randomly assigned to receive either self-directed (i.e., experimental) or facilitator-led (i.e., active control (AC)) VEGA.
Who Masked: Outcomes Assessor
Masking Description: The Research Assistant will be blinded to group allocation. The RA will be responsible for following-up with participants to make sure they've completed quantitative assessments (online survey) or, if participants choose to complete the surveys over the phone, the RA will complete them over the phone with the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Facilitator-Led VEGA (Active Comparator): Facilitator-led VEGA uses a group-based approach where participants complete the Violence, Evidence, Guidance, Action Project (VEGA) content as a virtual or face-to-face workshop. In this study, all workshops will be virtual to prevent social gathering during COVID-19.
  If a participant is randomized to this arm, the active control (AC) arm, they will be informed that they need to attend a facilitator-led VEGA session via virtual workshop format. The AC intervention will be facilitated via Zoom technology, by two trained facilitators with between 10 to 20 participants in each workshop (keeping the recommended 10:1 participant-to-facilitator ratio) and will last approximately 3 hours. The workshop approach is delivered by trained facilitators and is standardized via the use of a flexibly structured facilitator's guide. Facilitator-led VEGA will deliver material didactically with synchronous lecturing, use case-based role play, and include group-based polling.
  Interventions: Other: Violence, Evidence, Guidance, Action Project (VEGA) Education Intervention
- Self-Directed VEGA (Experimental): Self-directed VEGA uses an approach where participants complete the Violence, Evidence, Guidance, Action Project (VEGA) content online as a self-directed educational activity, at their own pace in a series of modules. Individuals will register to access the VEGA Educational Resources site. Participants have the option of completing the self-directed VEGA arm in either English or French as the VEGA Educational Resources site offers the content in French and English.
  If a participant is randomized to the experimental arm, they will be asked to complete the self-directed VEGA at their convenience, within one week of when they are informed they have been asked to complete the self-directed VEGA program. It will take approximately 3 hours for participants to complete all modules.
  Participants will read didactic material, complete case-based animated simulations, and complete individual multiple-choice questions with response feedback.
  Interventions: Other: Violence, Evidence, Guidance, Action Project (VEGA) Education Intervention

INTERVENTIONS:
Other: Violence, Evidence, Guidance, Action Project (VEGA) Education Intervention — VEGA is a novel education intervention that has the potential to improve the preparation of healthcare and social service providers (HHSPs) to be able to effectively recognize and respond to intimate partner violence (IPV) and related forms of family violence, including child maltreatment (CM), in their clinical encounters. VEGA was developed based on systematic reviews and consultation with individuals belonging to 22 national healthcare and social service organizations, including the Royal College of Physicians and Surgeons of Canada. VEGA follows a competency-based framework and a participatory, encounter-based curriculum that includes four learning modules: (a) the epidemiology of IPV and CM; (b) strategies for safely recognizing and responding to (i) IPV and (ii) CM; and (c) principles for ensuring safe clinical encounters for IPV and CM discussions.
  Other Names: VEGA Family Violence Education Resources

SUMMARY:
Prevention of child maltreatment (CM) remains a public health priority in Canada; approximately one-third of Canadians report exposure to at least one form of CM. Physicians play an important role in recognizing and responding to CM and its associated sequelae. However, increasing evidence indicates that physicians receive insufficient training related to recognizing and responding to CM. CM education is especially pertinent during the pediatric and psychiatry residency period but it remains unclear what the optimal approach is for preparing Canadian physicians with the knowledge and skills to effectively recognize and respond to CM. Those educational interventions that have been evaluated in medical education contexts have comparatively little emphasis on the complex overlap between IPV, children's exposure to IPV, and other forms of CM. The Violence, Evidence, Guidance, Action Project (VEGA) is a novel educational intervention that has the potential to improve the preparation of physicians to be able to effectively recognize and respond to CM in their clinical encounters and takes into account this complex overlap. The purpose of this study is to assess the acceptability and feasibility of a future randomized-controlled trial comparing two approaches to administering the VEGA intervention, facilitator-led or self-directed VEGA and whether/how these approaches can support residents' education.

The investigators hypothesize that there will be significant increases in preparedness, knowledge and skills, and self-efficacy to recognize and respond to CM in both the experimental and AC arms from Time 1 (baseline) to Time 2 (immediately after the intervention) and Time 1 (baseline) to Time 3 (3 month follow-up). The investigators also predict that these improvements will be slightly attenuated in the experimental arm. Qualitative data pertaining to perceived value and impact will corroborate the quantitative findings.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a resident at a Canadian University.
* Participant is fluent in written and spoken English.

Exclusion Criteria:

* Participant has previously accessed VEGA intervention materials.
* Participant is currently enrolled in or plans to enroll in any other educational intervention focused on family violence within the study time period (approximately next 3 months).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Residents Who Meet Eligibility Criteria | Through study completion, an average of 4 months
  The RC will track the number of residents who meet eligibility criteria, our aims are that we will recruit a total of 80 participants within 8 weeks, an average of 10 residents per week.
Number of Residents who Consent | Through study completion, an average of 4 months
  The RC will track the number of residents who consent to the study and agree to be randomized to either self-directed or facilitator-led VEGA education approaches, both overall and per week of recruitment. Our aim is that the proportion of residents who contact the research team about participation and who consent to randomization will be 75% or greater.
Number of Residents who Complete Assigned Intervention | Through study completion, an average of 4 months
  The RC will track the proportion of residents who are randomized and complete each arm, with completion consisting of reviewing all module content and the animated simulations in the case of self-directed VEGA and full attendance of the virtual workshop in the case of facilitator-led VEGA. Our goal is that the proportion of residents who are randomized and complete the assigned intervention will be 75% or greater for each arm. The acceptability of the facilitator-led and self-directed educational approaches as well as their value and impact will be determined via the coding of qualitative interview data from a sub-sample of participants.
Number of Residents who Complete Assessments | Through study completion, an average of 4 months
  The RC will track the feasibility of collecting trial outcome data (survey assessments) at Time 1, Time 2, and Time 3. Our goal is that the proportion of missing data for each time point will be less than 20%. Qualitative description will be used to expand and extend what we learn about acceptability and feasibility of implementing the associated research activities, we anticipate participants will not identify any fatal flaws related to the conduct of an RCT.

SECONDARY OUTCOMES:
Child Maltreatment Vignette Scale | Time 1 (one week before intervention), Time 2 (immediately after the intervention), Time 3 (3 month follow-up)
  Child Maltreatment Vignette scale (Pelletier et al., 2014; Pelletier & Knox, 2017) is a psychometrically validated measure of knowledge and skill accuracy related to recognizing and responding to child maltreatment. Respondents will be prompted to review 14 distinct analog vignettes that depict a range of signs and symptoms of possible CM exposure and asked if they suspect child maltreatment and if they would report to Child Welfare Services. Changes to the question wording and small changes to the wording of the scenarios were made to align the measure with the Canadian context. A mean "knowledge and skill accuracy" score will be produced for analysis, with higher scores indicative of greater knowledge and skill accuracy related to CM. In a future RCT, this would be one of the primary outcomes of interest since this is a robust measure of knowledge and skills related to CM.
Child Maltreatment Knowledge and Skills Questions (Developed by VEGA Team) | Time 1 (one week before intervention), Time 2 (immediately after the intervention), Time 3 (3 month follow-up)
  Participants will be asked a series of questions about their knowledge and skills related to recognizing and responding to child maltreatment. These were developed by the VEGA training research team to capture specific aspects of child maltreatment knowledge directly addressed in the VEGA intervention and which are outside the scope of the child maltreatment vignette scale. The questions ask about the following topics (and more not mentioned here): parental/family risk factors for family violence, what future outcomes are associated with child maltreatment, other possible signs of child abuse, and principles for good documentation and providing ongoing care to children experiencing maltreatment. Including this measure in our study will allow us to make cross sample comparisons.
The Physician Readiness to Manage Intimate Partner Violence Survey: Preparedness Subscale | Time 1 (one week before intervention), Time 3 (3 month follow-up)
  The Physician Readiness to Manage Intimate Partner Violence Survey (PREMIS) is a 67-item self-report tool that was developed to assess physician management of intimate partner violence across 10 subscales (Short et al.,2006; Connor et al., 2011). The preparedness subscale of PREMIS asks respondents to indicate the extent to which they feel prepared to address various aspects of IPV recognition and response when working with their clients across 10 items, including asking appropriate questions about IPV and responding to IPV disclosures. Response options are on a 7-item Likert type scale ranging from "Not prepared" (1) to "Quite Well Prepared" (7) and items are averaged to generate a mean score for practitioner preparedness, with higher scores indicative of greater perceived preparedness to recognize and respond to IPV. All items will be changed to be related to child maltreatment instead of IPV, several items were dropped as they are not relevant in the case of CM.
Mandatory Reporting Self-Efficacy Scale (MRSES) | Time 1 (one week before intervention), Time 2 (immediately after the intervention), Time 3 (3 month follow-up)
  The MRSES is a 7-item self-report measure that asks respondents to indicate the extent to which they perceive their ability to implement a series of behaviours related to mandatory reporting of CM (Ayling, 2019). Informed by Bandura's self-efficacy theory and recommendations for self-efficacy scales (Bandura, 2006), response options are anchored on a scale from 0 to 100 with: "cannot do at all (0)"; moderately can do (50)"; and "highly certain can do (100)." A total score is generated by summing items across the scale for each participant, with higher scores indicative of greater self-efficacy related to recognizing and reporting suspected CM. We anticipate that this measure will be a key mediator of interest in a future definitive RCT given that across provincial and territorial jurisdictions in Canada (including Ontario), a suspicion of CM meets the threshold for a report to child protection authorities (Dubowitz, 2014; Mathews and Kenny, 2008).
Brief Individual Readiness for Change Scale (BIRCS) | Time 1 (one week before intervention)
  The BIRCS scale is a 5-item readiness for change tool (Goldman, 2009). The scale's purpose is to screen for practitioners' readiness for change, in other words their receptivity to learning and applying new evidence-based research practices. For the purpose of this study, the items were adapted to assess provider's readiness to recognize and respond to all forms of child maltreatment (CM) in their clinical encounters. Response options range from '0' Strongly Disagree to '4' Strongly Agree. Two items were added, "I believe recognizing and responding to child maltreatment in my practice improves outcomes for my clients," and "I am motivated to learn about child maltreatment" to capture other aspects of residents' readiness to learn about CM and their belief's about how this will impact their practice.
Achievement Goals for Work Domain (AGWD) | Time 1 (one week before intervention)
  The Achievement Goals for Work Domain (AGWD) scale is a 23-item, psychometrically validated measure of work-related achievement goals that map onto the four goal orientations described by Achievement Goal Theory (Daniels & Daniels, 2018; Baranik et al., 2007). Respondents are asked to indicate their agreement with 23 statements, response options range from '1' strongly disagree to '7' strongly agree and responses are summed to generate a total score for each subscale corresponding to each type of goal orientation; higher scores are more indicative of the respondent's affinity to that goal orientation. In this study, they will be asked about their achievement goals for residency.

OTHER OUTCOMES:
Demographics | Pre-Intervention
  Sociodemographic characteristics will be collected for all participants who are screened for the study, whether they are ineligible or eligible. These will include their age, their program (psychiatry or pediatrics), their sex at birth and their self-identified gender.
Previous Training in Child Maltreatment | Time 1 (one week before intervention)
  Participants will be asked questions to gauge their previous education or training in various areas of CM. Participants will be given a definition of CM and asked in what areas they have received education or training related to CM, in what environment(s) they have learned about CM, and in which of these environments they have learned the most.
Thoughts and Beliefs about Recognizing and Responding to CM in Professional Roles | Time 1 (one week before intervention)
  Participants will be asked to rate their agreement with two statements about how much they believe (1) recognizing and (2) responding to CM is a part of their professional role. In qualitative interviews we will ask participants how often they believe they will encounter family violence in their future practice (how relevant it is to their future professional role as a psychiatrist or pediatrician), the purpose of these questions is to gauge this in our entire sample.
Satisfaction with VEGA Training | Time 2 (immediately after the intervention)
  Participants will complete a series of multiple choice and short-answer questions asking what they thought about the VEGA training. These questions will apply to all participants whether they completed self-directed or facilitator-led VEGA. Questions will include whether they believe the intended learning outcomes were achieved, what they thought of the instructional materials and educational scenarios, and how they would rate the usefulness of VEGA.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Kimber, PhD, MSW, RSW, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Requests for data for analyses (e.g. by Research Team Members, graduate trainees) will be managed by the research coordinator and overseen by the PI, including Dr. Melissa Kimber. This will not include identifying information of participants, only de-identified data would be shared.

REFERENCES:
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Pelletier HL, Knox M. Incorporating Child Maltreatment Training into Medical School Curricula. J Child Adolesc Trauma. 2017;10(3):267-274. doi: 10.1007/s40653-016-0096-x. Epub 2016 May 12. PMID 29026450
- [Background] Connor PD, Nouer SS, Mackey ST, Tipton NG, Lloyd AK. Psychometric properties of an intimate partner violence tool for health care students. J Interpers Violence. 2011 Mar;26(5):1012-35. doi: 10.1177/0886260510365872. Epub 2010 Jun 28. PMID 20587479
- [Background] Short LM, Alpert E, Harris JM Jr, Surprenant ZJ. A tool for measuring physician readiness to manage intimate partner violence. Am J Prev Med. 2006 Feb;30(2):173-180. doi: 10.1016/j.amepre.2005.10.009. PMID 16459217
- [Background] Mathews B, Kenny MC. Mandatory reporting legislation in the United States, Canada, and Australia: a cross-jurisdictional review of key features, differences, and issues. Child Maltreat. 2008 Feb;13(1):50-63. doi: 10.1177/1077559507310613. PMID 18174348
- [Background] Daniels L, Daniels V. Internal medicine residents' achievement goals and efficacy, emotions, and assessments. Can Med Educ J. 2018 Nov 12;9(4):e59-e68. eCollection 2018 Nov. PMID 30498544
- [Background] MacMillan HL, Kimber M, Stewart DE. Intimate Partner Violence: Recognizing and Responding Safely. JAMA. 2020 Sep 22;324(12):1201-1202. doi: 10.1001/jama.2020.11322. No abstract available. PMID 32960228
- [Background] Stewart DE, MacMillan H, Kimber M. Recognizing and Responding to Intimate Partner Violence: An Update. Can J Psychiatry. 2021 Jan;66(1):71-106. doi: 10.1177/0706743720939676. Epub 2020 Aug 10. No abstract available. PMID 32777936
- [Background] Kimber M, McTavish JR, Couturier J, Le Grange D, Lock J, MacMillan HL. Identifying and responding to child maltreatment when delivering family-based treatment-A qualitative study. Int J Eat Disord. 2019 Mar;52(3):292-298. doi: 10.1002/eat.23036. Epub 2019 Feb 6. PMID 30729594
- [Background] Kimber M, McTavish JR, Luo C, Couturier J, Dimitropoulos G, MacMillan H. Mandatory reporting of child maltreatment when delivering family-based treatment for eating disorders: A framework analysis of practitioner experiences. Child Abuse Negl. 2019 Feb;88:118-128. doi: 10.1016/j.chiabu.2018.11.010. Epub 2018 Nov 23. PMID 30476720
- [Background] McTavish JR, Kimber M, Devries K, Colombini M, MacGregor JCD, Wathen CN, Agarwal A, MacMillan HL. Mandated reporters' experiences with reporting child maltreatment: a meta-synthesis of qualitative studies. BMJ Open. 2017 Oct 16;7(10):e013942. doi: 10.1136/bmjopen-2016-013942. PMID 29042370
- [Background] Alnasser Y, Albijadi A, Abdullah W, Aldabeeb D, Alomair A, Alsaddiqi S, Alsalloum Y. Child maltreatment between knowledge, attitude and beliefs among Saudi pediatricians, pediatric residency trainees and medical students. Ann Med Surg (Lond). 2017 Feb 21;16:7-13. doi: 10.1016/j.amsu.2017.02.008. eCollection 2017 Apr. PMID 28275426
- [Background] Flaherty EG, Sege R, Price LL, Christoffel KK, Norton DP, O'Connor KG. Pediatrician characteristics associated with child abuse identification and reporting: results from a national survey of pediatricians. Child Maltreat. 2006 Nov;11(4):361-9. doi: 10.1177/1077559506292287. PMID 17043321
- [Background] Flaherty EG, Sege R, Binns HJ, Mattson CL, Christoffel KK. Health care providers' experience reporting child abuse in the primary care setting. Pediatric Practice Research Group. Arch Pediatr Adolesc Med. 2000 May;154(5):489-93. doi: 10.1001/archpedi.154.5.489. PMID 10807301
- [Background] Regnaut O, Jeu-Steenhouwer M, Manaouil C, Gignon M. Risk factors for child abuse: levels of knowledge and difficulties in family medicine. A mixed method study. BMC Res Notes. 2015 Oct 30;8:620. doi: 10.1186/s13104-015-1607-9. PMID 26514128
- [Background] Flaherty EG, Sege R. Barriers to physician identification and reporting of child abuse. Pediatr Ann. 2005 May;34(5):349-56. doi: 10.3928/0090-4481-20050501-08. PMID 15948346
- [Background] Norman GR, Sloan JA, Wyrwich KW. The truly remarkable universality of half a standard deviation: confirmation through another look. Expert Rev Pharmacoecon Outcomes Res. 2004 Oct;4(5):581-5. doi: 10.1586/14737167.4.5.581. PMID 19807551
- [Background] Crowe M, Inder M, Porter R. Conducting qualitative research in mental health: Thematic and content analyses. Aust N Z J Psychiatry. 2015 Jul;49(7):616-23. doi: 10.1177/0004867415582053. Epub 2015 Apr 21. PMID 25900973
- [Background] Guetterman TC, Fetters MD, Creswell JW. Integrating Quantitative and Qualitative Results in Health Science Mixed Methods Research Through Joint Displays. Ann Fam Med. 2015 Nov;13(6):554-61. doi: 10.1370/afm.1865. PMID 26553895
- [Background] Brown DS, Fang X, Florence CS. Medical costs attributable to child maltreatment a systematic review of short- and long-term effects. Am J Prev Med. 2011 Dec;41(6):627-35. doi: 10.1016/j.amepre.2011.08.013. PMID 22099241
- [Background] Afifi TO, MacMillan HL, Boyle M, Taillieu T, Cheung K, Sareen J. Child abuse and mental disorders in Canada. CMAJ. 2014 Jun 10;186(9):E324-32. doi: 10.1503/cmaj.131792. Epub 2014 Apr 22. PMID 24756625
- [Background] Bair-Merritt MH, Blackstone M, Feudtner C. Physical health outcomes of childhood exposure to intimate partner violence: a systematic review. Pediatrics. 2006 Feb;117(2):e278-90. doi: 10.1542/peds.2005-1473. PMID 16452335
- [Background] Caslini M, Bartoli F, Crocamo C, Dakanalis A, Clerici M, Carra G. Disentangling the Association Between Child Abuse and Eating Disorders: A Systematic Review and Meta-Analysis. Psychosom Med. 2016 Jan;78(1):79-90. doi: 10.1097/PSY.0000000000000233. PMID 26461853
- [Background] Chen LP, Murad MH, Paras ML, Colbenson KM, Sattler AL, Goranson EN, Elamin MB, Seime RJ, Shinozaki G, Prokop LJ, Zirakzadeh A. Sexual abuse and lifetime diagnosis of psychiatric disorders: systematic review and meta-analysis. Mayo Clin Proc. 2010 Jul;85(7):618-29. doi: 10.4065/mcp.2009.0583. Epub 2010 May 10. PMID 20458101
- [Background] Danese A, Tan M. Childhood maltreatment and obesity: systematic review and meta-analysis. Mol Psychiatry. 2014 May;19(5):544-54. doi: 10.1038/mp.2013.54. Epub 2013 May 21. PMID 23689533
- [Background] Kimber M, McTavish JR, Couturier J, Boven A, Gill S, Dimitropoulos G, MacMillan HL. Consequences of child emotional abuse, emotional neglect and exposure to intimate partner violence for eating disorders: a systematic critical review. BMC Psychol. 2017 Sep 22;5(1):33. doi: 10.1186/s40359-017-0202-3. PMID 28938897
- [Background] Pignatelli AM, Wampers M, Loriedo C, Biondi M, Vanderlinden J. Childhood neglect in eating disorders: A systematic review and meta-analysis. J Trauma Dissociation. 2017 Jan-Feb;18(1):100-115. doi: 10.1080/15299732.2016.1198951. Epub 2016 Jun 9. PMID 27282982
- [Background] Lindert J, von Ehrenstein OS, Grashow R, Gal G, Braehler E, Weisskopf MG. Sexual and physical abuse in childhood is associated with depression and anxiety over the life course: systematic review and meta-analysis. Int J Public Health. 2014 Apr;59(2):359-72. doi: 10.1007/s00038-013-0519-5. PMID 24122075
- [Background] Norman RE, Byambaa M, De R, Butchart A, Scott J, Vos T. The long-term health consequences of child physical abuse, emotional abuse, and neglect: a systematic review and meta-analysis. PLoS Med. 2012;9(11):e1001349. doi: 10.1371/journal.pmed.1001349. Epub 2012 Nov 27. PMID 23209385
- [Background] Suglia SF, Sapra KJ, Koenen KC. Violence and cardiovascular health: a systematic review. Am J Prev Med. 2015 Feb;48(2):205-212. doi: 10.1016/j.amepre.2014.09.013. PMID 25599905
- [Background] Beynon CE, Gutmanis IA, Tutty LM, Wathen CN, MacMillan HL. Why physicians and nurses ask (or don't) about partner violence: a qualitative analysis. BMC Public Health. 2012 Jun 21;12:473. doi: 10.1186/1471-2458-12-473. PMID 22721371
- [Background] Inanici SY, Celik E, Hidiroglu S, Ozdemir M, Inanici MA. Factors associated with physicians' assessment and management of child abuse and neglect: A mixed method study. J Forensic Leg Med. 2020 Jul;73:101972. doi: 10.1016/j.jflm.2020.101972. Epub 2020 May 30. PMID 32658746
- [Background] Flaherty EG, Sege R, Mattson CL, Binns HJ. Assessment of suspicion of abuse in the primary care setting. Ambul Pediatr. 2002 Mar-Apr;2(2):120-6. doi: 10.1367/1539-4409(2002)0022.0.co;2. PMID 11926843
- [Background] Kuruppu J, McKibbin G, Humphreys C, Hegarty K. Tipping the Scales: Factors Influencing the Decision to Report Child Maltreatment in Primary Care. Trauma Violence Abuse. 2020 Jul;21(3):427-438. doi: 10.1177/1524838020915581. Epub 2020 Apr 7. PMID 32254001
- [Background] Lewis NV, Feder GS, Howarth E, Szilassy E, McTavish JR, MacMillan HL, Wathen N. Identification and initial response to children's exposure to intimate partner violence: a qualitative synthesis of the perspectives of children, mothers and professionals. BMJ Open. 2018 Apr 28;8(4):e019761. doi: 10.1136/bmjopen-2017-019761. PMID 29705757
- [Background] McTavish JR, Kimber M, Devries K, Colombini M, MacGregor JCD, Wathen N, MacMillan HL. Children's and caregivers' perspectives about mandatory reporting of child maltreatment: a meta-synthesis of qualitative studies. BMJ Open. 2019 Apr 4;9(4):e025741. doi: 10.1136/bmjopen-2018-025741. PMID 30948587
- [Background] Divakar U, Nazeha N, Posadzki P, Jarbrink K, Bajpai R, Ho AHY, Campbell J, Feder G, Car J. Digital Education of Health Professionals on the Management of Domestic Violence: Systematic Review and Meta-Analysis by the Digital Health Education Collaboration. J Med Internet Res. 2019 May 23;21(5):e13868. doi: 10.2196/13868. PMID 31124462
- [Background] Sawyer S, Coles J, Williams A, Williams B. A systematic review of intimate partner violence educational interventions delivered to allied health care practitioners. Med Educ. 2016 Nov;50(11):1107-1121. doi: 10.1111/medu.13108. PMID 27762036
- [Background] Turner W, Hester M, Broad J, Szilassy E, Feder G, Drinkwater J, Firth A, Stanley N. Interventions to Improve the Response of Professionals to Children Exposed to Domestic Violence and Abuse: A Systematic Review. Child Abuse Rev. 2017 Jan-Feb;26(1):19-39. doi: 10.1002/car.2385. Epub 2015 Jun 29. PMID 28392674
- [Background] Zaher E, Keogh K, Ratnapalan S. Effect of domestic violence training: systematic review of randomized controlled trials. Can Fam Physician. 2014 Jul;60(7):618-24, e340-7. PMID 25022633
- [Background] Hamberger LK. Preparing the next generation of physicians: medical school and residency-based intimate partner violence curriculum and evaluation. Trauma Violence Abuse. 2007 Apr;8(2):214-25. doi: 10.1177/1524838007301163. PMID 17545575
- [Background] Vaismoradi M, Turunen H, Bondas T. Content analysis and thematic analysis: Implications for conducting a qualitative descriptive study. Nurs Health Sci. 2013 Sep;15(3):398-405. doi: 10.1111/nhs.12048. Epub 2013 Mar 11. PMID 23480423
- [Background] Adams NE. Bloom's taxonomy of cognitive learning objectives. J Med Libr Assoc. 2015 Jul;103(3):152-3. doi: 10.3163/1536-5050.103.3.010. PMID 26213509
- [Background] Armson H, Elmslie T, Roder S, Wakefield J. Is the Cognitive Complexity of Commitment-to-Change Statements Associated With Change in Clinical Practice? An Application of Bloom's Taxonomy. J Contin Educ Health Prof. 2015 Summer;35(3):166-75. doi: 10.1002/chp.21303. PMID 26378422
- [Background] Shannon S. Educational objectives for CME programmes. Lancet. 2003 Apr 12;361(9365):1308. doi: 10.1016/S0140-6736(03)13020-6. No abstract available. PMID 12699998
- [Background] Su WM, Osisek PJ. The Revised Bloom's Taxonomy: implications for educating nurses. J Contin Educ Nurs. 2011 Jul;42(7):321-7. doi: 10.3928/00220124-20110621-05. PMID 21707023
- [Background] Larsen DP, Butler AC, Roediger HL 3rd. Test-enhanced learning in medical education. Med Educ. 2008 Oct;42(10):959-66. doi: 10.1111/j.1365-2923.2008.03124.x. PMID 18823514
- [Background] McLean SF. Case-Based Learning and its Application in Medical and Health-Care Fields: A Review of Worldwide Literature. J Med Educ Curric Dev. 2016 Apr 27;3:JMECD.S20377. doi: 10.4137/JMECD.S20377. eCollection 2016 Jan-Dec. PMID 29349306
- [Background] Jordan J, Jalali A, Clarke S, Dyne P, Spector T, Coates W. Asynchronous vs didactic education: it's too early to throw in the towel on tradition. BMC Med Educ. 2013 Aug 8;13:105. doi: 10.1186/1472-6920-13-105. PMID 23927420
- [Background] Ericsson KA. Deliberate practice and acquisition of expert performance: a general overview. Acad Emerg Med. 2008 Nov;15(11):988-94. doi: 10.1111/j.1553-2712.2008.00227.x. Epub 2008 Sep 5. PMID 18778378
- [Background] Akl EA, Pretorius RW, Sackett K, Erdley WS, Bhoopathi PS, Alfarah Z, Schunemann HJ. The effect of educational games on medical students' learning outcomes: a systematic review: BEME Guide No 14. Med Teach. 2010 Jan;32(1):16-27. doi: 10.3109/01421590903473969. PMID 20095770
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Murad MH, Coto-Yglesias F, Varkey P, Prokop LJ, Murad AL. The effectiveness of self-directed learning in health professions education: a systematic review. Med Educ. 2010 Nov;44(11):1057-68. doi: 10.1111/j.1365-2923.2010.03750.x. PMID 20946476
- [Background] Cook DA, Levinson AJ, Garside S, Dupras DM, Erwin PJ, Montori VM. Internet-based learning in the health professions: a meta-analysis. JAMA. 2008 Sep 10;300(10):1181-96. doi: 10.1001/jama.300.10.1181. PMID 18780847
- [Background] Norman G. RCT = results confounded and trivial: the perils of grand educational experiments. Med Educ. 2003 Jul;37(7):582-4. doi: 10.1046/j.1365-2923.2003.01586.x. No abstract available. PMID 12834412
- [Background] Norman G. The end of educational science? Adv Health Sci Educ Theory Pract. 2008 Nov;13(4):385-9. doi: 10.1007/s10459-008-9139-x. Epub 2008 Oct 21. No abstract available. PMID 18941917
- [Background] Sullivan GM. Getting off the "gold standard": randomized controlled trials and education research. J Grad Med Educ. 2011 Sep;3(3):285-9. doi: 10.4300/JGME-D-11-00147.1. No abstract available. PMID 22942950
- [Derived] Kimber M, Baker-Sullivan E, Stewart DE, Vanstone M. Improving Health Professional Recognition and Response to Child Maltreatment and Intimate Partner Violence: Protocol for Two Mixed Methods Pilot Randomized Controlled Trials. JMIR Res Protoc. 2024 Mar 21;13:e50864. doi: 10.2196/50864. PMID 38512307
- See also: This is the VEGA Project website, where the public can access VEGA Family Violence Education Resources. More information can be found here about the development of VEGA. — https://vegaproject.mcmaster.ca/